CLINICAL TRIAL: NCT02764151
Title: A PHASE 1 DOSE ESCALATION STUDY EVALUATING THE SAFETY AND TOLERABILITY OF PF-06840003 IN PATIENTS WITH MALIGNANT GLIOMAS
Brief Title: First in Patient Study for PF-06840003 in Malignant Gliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to prematurely terminate the study and not to pursue marketing approval for the indication of malignant glioma.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0591001
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Oligodendroglioma; Astrocytoma; Malignant Glioma
Keywords: GBM; malignant glioma; glioma; anaplastic glioma; astrocytoma; IDO; IDO1; PF-06840003
MeSH Terms: conditions — Oligodendroglioma; Astrocytoma; Glioma | interventions — PF-06840003

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-06840003 (Experimental): Daily Oral PF-06840003
  Interventions: Drug: PF-06840003

INTERVENTIONS:
Drug: PF-06840003 — Daily Oral PF-06840003

SUMMARY:
This study will evaluate the safety and tolerability of increasing doses of PF-06840003 in patients with malignant gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of WHO Grade IV glioblastoma or WHO Grade III anaplastic gliomas
* For patients with Grade IV GBM, recurrent disease at the time of the first or second recurrence or progression. For patients with Grade III anaplastic gliomas, recurrent disease at the time of at least a first recurrence but no more than a fourth recurrence or progression
* Karnofsky performance score greater than or equal to 70%
* Adequate bone marrow, kidney and liver function

Exclusion Criteria:

* History of CNS bleeding within 6 months of registration
* Previous anti-angiogenics or anti-vascular endothelial growth factor within 12 months of registration
* Requires treatment with high dose systemic corticosteroids defined as >2 mg/day
* Radiation therapy within 12 weeks of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Clinical & Translational Research Center, Los Angeles, California
  - UCLA Oncology Center, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - CUMC Research Pharmacy, New York, New York
  - Columbia Doctors Tarrytown, Tarrytown, New York
  - Duke Cancer Center, Durham, North Carolina
  - Duke University Medical Center, Duke Cancer Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Reardon DA, Desjardins A, Rixe O, Cloughesy T, Alekar S, Williams JH, Li R, Taylor CT, Lassman AB. A phase 1 study of PF-06840003, an oral indoleamine 2,3-dioxygenase 1 (IDO1) inhibitor in patients with recurrent malignant glioma. Invest New Drugs. 2020 Dec;38(6):1784-1795. doi: 10.1007/s10637-020-00950-1. Epub 2020 May 20. PMID 32436060
- [Derived] Gomes B, Driessens G, Bartlett D, Cai D, Cauwenberghs S, Crosignani S, Dalvie D, Denies S, Dillon CP, Fantin VR, Guo J, Letellier MC, Li W, Maegley K, Marillier R, Miller N, Pirson R, Rabolli V, Ray C, Streiner N, Torti VR, Tsaparikos K, Van den Eynde BJ, Wythes M, Yao LC, Zheng X, Tumang J, Kraus M. Characterization of the Selective Indoleamine 2,3-Dioxygenase-1 (IDO1) Catalytic Inhibitor EOS200271/PF-06840003 Supports IDO1 as a Critical Resistance Mechanism to PD-(L)1 Blockade Therapy. Mol Cancer Ther. 2018 Dec;17(12):2530-2542. doi: 10.1158/1535-7163.MCT-17-1104. Epub 2018 Sep 19. PMID 30232146
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0591001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After reviewing efficacy, safety, PK and PD of all available data from enrolled patients, the Sponsor decided to prematurely terminate the study and not to pursue marketing approval for PF-06840003 in the indication of malignant glioma. Part 2 of the study was not initiated.
Groups:
- PF-06840003 125 MG QD: PF-06840003 (formulated 125 mg tablets) was administered orally at 125 mg once daily (QD) for 28-day cycles.
- PF-06840003 250 MG QD: PF-06840003 (formulated 125 mg tablets) was administered orally at 250 mg QD for 28-day cycles.
- PF-06840003 250 MG BID: PF-06840003 (formulated 125 mg tablets) was administered orally at 250 mg twice daily (BID) for 28-day cycles.
- PF-06840003 500 MG BID: PF-06840003 (formulated 125 mg tablets) was administered orally at 500 mg BID for 28-day cycles.
Period: Overall Study
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Started | 2 | 4 | 3 | 8
Completed | 2 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 3
Not completed — Subject refused further follow-up | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All Part 1 enrolled participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID | Total
Number analyzed (Participants) | 2 | 4 | 3 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (19.1) | 51.8 (14.5) | 49.3 (12.1) | 58.1 (14.6) | 53.5 (14.1)
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 1 | 2 | 1 | 1 | 5
  45-64 Years | 1 | 1 | 2 | 3 | 7
  >=65 Years | 0 | 1 | 0 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 3 | 5
  Male | 1 | 4 | 2 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 4 | 3 | 7 | 16
  Asian | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) [Part 1]
Description: DLTs: Any of the following adverse events (AE) occurring in the first cycle of treatment, unless there is a clear alternative explanation. Hematologic: Grade (Gr) 4 neutropenia lasting >=5 days; febrile neutropenia; Gr>=3 neutropenic with infection; Gr>=3 thrombocytopenia with bleeding; Gr 4 thrombocytopenia. Non-Hematologic: Any toxicity attributable to PF-06840003 that resulted in administration of less than 80% of the planned doses during Cycle 1; Gr 4 non-hematologic AE; Gr 3 AE lasting >7 days despite optimal supportive care; Gr 3 central nervous system (CNS) AE regardless of duration; Gr 3 QTc prolongation (QTc >500 milliseconds) (a DLT only if persisting after correction of any reversible causes); Concurrent aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3*upper limit of normal (ULN) and total bilirubin >2*ULN.
Time Frame: Baseline to Day 28
Population: All Part 1 enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Participants | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) [Part 1]
Description: An AE was any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were those with initial onset or increasing in severity after the first dose of study treatment.
Time Frame: Baseline up to 1 year
Population: All Part 1 enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Participants
  All-causality TEAEs | 2 | 4 | 3 | 8
  Treatment-related TEAEs | 1 | 4 | 2 | 7

3. Primary Outcome: Number of Participants With TEAEs by Severity (as Graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Event [CTCAE] Version 4.03) [Part 1]
Description: Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. AEs were graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03: Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: Baseline up to 1 year
Population: All Part 1 enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Participants
  Grade 3 or 4 | 0 | 1 | 1 | 2
  Grade 5 | 0 | 0 | 0 | 0

4. Secondary Outcome: Objective Response Rate (ORR) [Part 1]
Description: Objective response rate (ORR), defined as the percentage of patients achieving complete response (CR) or partial response (PR) as assessed by Macdonald criteria: CR: complete disappearance of all enhancing measurable and non-measurable disease on consecutive MRI at least 4 weeks apart, off steroid, sustained for at least 4 weeks; PR: >=50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks.
Time Frame: Weeks 8, 16, and 24
Population: The analysis population included all the participants enrolled.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Percentage of Participants
  Week 8 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94]
  Week 16 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94]
  Week 24 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94]

5. Secondary Outcome: Disease Control Rate (DCR) Based on the Immunotherapy Response Assessment for Neuro-Oncology (iRANO) Criteria [Part 1]
Description: Disease control rate (DCR) was defined as the percentage of patients achieving CR, PR, or stable disease (SD). Overall DCR was based on iRANO criteria: CR: complete disappearance of all enhancing measurable and non-measurable disease on consecutive MRI at least 4 weeks apart, off steroid, sustained for at least 4 weeks; PR: >=50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; SD: does not qualify for CR, PR, or progression disease, and stable clinically.
Time Frame: Weeks 8, 16, and 24
Population: The analysis population included all the participants enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
percentage of participants
  Week 8 | 50.0 [1.26 to 98.74] | 50.0 [6.76 to 93.24] | 33.3 [0.84 to 90.57] | 25.0 [3.19 to 65.09]
  Week 16 | 50.0 [1.26 to 98.74] | 0.0 [0.00 to 60.24] | 66.7 [9.43 to 99.16] | 25.0 [3.19 to 65.09]
  Week 24 | 0.0 [0.00 to 84.19] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 70.76] | 25.0 [3.19 to 65.09]

6. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities by Severity (as Graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Event [CTCAE] Version 4.03) [Part 1]
Description: Following parameters were analyzed for hematology laboratory test: hemoglobin, platelets, white blood cell (WBC), absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils, and absolute basophils. Laboratory abnormalities were graded per NCI CTCAE version 4.03 and those with at least 1 participant are presented here.
Time Frame: Baseline up to 1 year
Population: All Part 1 enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Participants
  Anemia, Grade 0 | 1 | 2 | 0 | 2
  Anemia, Grade 1 | 0 | 2 | 3 | 6
  Anemia, Grade 2 | 1 | 0 | 0 | 0
  Hemoglobin increased, Grade 0 | 2 | 4 | 3 | 8
  Lymphocyte count increased, Grade 0 | 2 | 4 | 3 | 8
  Lymphopenia, Grade 0 | 1 | 2 | 1 | 5
  Lymphopenia, Grade 1 | 1 | 1 | 0 | 1
  Lymphopenia, Grade 2 | 0 | 1 | 1 | 0
  Lymphopenia, Grade 3 | 0 | 0 | 1 | 2
  Neutrophils (absolute), Grade 0 | 1 | 3 | 2 | 7
  Neutrophils (absolute), Grade 1 | 1 | 1 | 0 | 1
  Neutrophils (absolute), Grade 2 | 0 | 0 | 1 | 0
  Platelets, Grade 0 | 2 | 2 | 3 | 5
  Platelets, Grade 1 | 0 | 2 | 0 | 3
  WBC, Grade 0 | 2 | 3 | 1 | 6
  WBC, Grade 1 | 0 | 1 | 1 | 1
  WBC, Grade 2 | 0 | 0 | 1 | 1

7. Secondary Outcome: Number of Participants With Chemistries Laboratory Abnormalities by Severity (as Graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Event [CTCAE] Version 4.03) [Part 1]
Description: Following parameters were analyzed for chemistry laboratory test: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), alkaline phosphatase, sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen (BUN) or urea, creatinine, uric acid, glucose (non-fasted), albumin, and phosphorous or phosphate. Laboratory abnormalities were graded per NCI CTCAE version 4.03 and those with at least 1 participant are presented here.
Time Frame: Baseline up to 1 year
Population: All Part 1 enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Participants
  ALT, Grade 0 | 2 | 2 | 3 | 7
  ALT, Grade 1 | 0 | 1 | 0 | 0
  ALT, Grade 3 | 0 | 1 | 0 | 0
  ALT, Grade 4 | 0 | 0 | 0 | 1
  Alkaline phosphatase, Grade 0 | 2 | 3 | 3 | 6
  Alkaline phosphatase, Grade 1 | 0 | 1 | 0 | 2
  AST, Grade 0 | 2 | 3 | 3 | 7
  AST, Grade 2 | 0 | 1 | 0 | 0
  AST, Grade 4 | 0 | 0 | 0 | 1
  Bilirubin (total), Grade 0 | 2 | 4 | 3 | 8
  Creatinine, Grade 0 | 0 | 0 | 1 | 0
  Creatinine, Grade 1 | 2 | 4 | 2 | 7
  Creatinine, Grade 2 | 0 | 0 | 0 | 1
  Hypercalcemia, Grade 0 | 1 | 4 | 3 | 8
  Hypercalcemia, Grade 1 | 1 | 0 | 0 | 0
  Hyperglycemia, Grade 0 | 1 | 0 | 3 | 1
  Hyperglycemia, Grade 1 | 1 | 4 | 0 | 4
  Hyperglycemia, Grade 2 | 0 | 0 | 0 | 2
  Hyperglycemia, Grade 3 | 0 | 0 | 0 | 1
  Hyperkalemia, Grade 0 | 2 | 4 | 3 | 7
  Hyperkalemia, Grade 3 | 0 | 0 | 0 | 1
  Hypermagnesemia, Grade 0 | 2 | 4 | 3 | 7
  Hypermagnesemia, Grade 1 | 0 | 0 | 0 | 1
  Hypernatremia, Grade 0 | 2 | 4 | 3 | 7
  Hypernatremia, Grade 1 | 0 | 0 | 0 | 1
  Hypoalbuminemia, Grade 0 | 2 | 3 | 3 | 5
  Hypoalbuminemia, Grade 1 | 0 | 1 | 0 | 2
  Hypoalbuminemia, Grade 2 | 0 | 0 | 0 | 1
  Hypocalcemia, Grade 0 | 2 | 3 | 0 | 6
  Hypocalcemia, Grade 1 | 0 | 1 | 3 | 1
  Hypocalcemia, Grade 2 | 0 | 0 | 0 | 1
  Hypoglycemia, Grade 0 | 2 | 3 | 3 | 8
  Hypoglycemia, Grade 1 | 0 | 1 | 0 | 0
  Hypokalemia, Grade 0 | 2 | 4 | 1 | 4
  Hypokalemia, Grade 1 | 0 | 0 | 2 | 4
  Hypomagnesemia, Grade 0 | 2 | 4 | 2 | 8
  Hypomagnesemia, Grade 1 | 0 | 0 | 1 | 0
  Hyponatremia, Grade 0 | 2 | 4 | 1 | 7
  Hyponatremia, Grade 1 | 0 | 0 | 1 | 1
  Hyponatremia, Grade 3 | 0 | 0 | 1 | 0
  Hypophosphatemia, Grade 0 | 2 | 4 | 3 | 6
  Hypophosphatemia, Grade 2 | 0 | 0 | 0 | 2

8. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs [Part 1]
Description: Vital signs included measurements of blood pressure and temperature (oral, tympanic, temporal or axillary). The investigator judged any clinically significant vital signs findings.
Time Frame: Baseline up to 1 year
Population: All Part 1 enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Single Dose: Maximum Observed Plasma Concentration (Cmax) of PF-06840002 and PF-06840001 [Part 1]
Description: Cmax of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) were observed directly from data.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: The analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
nanograms per milliliter (ng/mL)
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 580.5 (468-693). | 775.0 (37) | 1135 (6) | 1407 (23)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 991.0 (792-1190). | 1309 (28) | 1763 (8) | 2286 (20)

10. Secondary Outcome: Single Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06840002 and PF-06840001 [Part 1]
Description: Tmax of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) were observed directly from data as time of first occurence.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: as for outcome 9
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
hour (hr)
  PF-06840002 | 1.58 [1.00 to 2.15] | 1.51 [1.00 to 2.08] | 1.95 [1.00 to 2.05] | 3.02 [1.00 to 4.05]
  PF-06840001 | 2.50 [1.00 to 4.00] | 2.05 [1.00 to 2.13] | 2.05 [1.95 to 4.00] | 3.98 [1.00 to 4.05]

11. Secondary Outcome: Single Dose: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PF-06840002 and PF-06840001 [Part 1]
Description: AUClast of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by linear/log trapezoidal method.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
nanogram*hour per milliliter (ng*hr/mL)
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 3155 (2450-3860). | 4517 (80) | 13340 (21) | 17720 (78)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 6250 (5790-6710). | 7626 (66) | 21670 (24) | 28250 (71)

12. Secondary Outcome: Single Dose: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06840002 and PF-06840001 [Part 1]
Description: AUCtau of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by linear/log trapezoidal method.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
nanogram*hour per milliliter (ng*hr/mL)
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 3380 (2900-3860). | 5356 (60) | 7606 (11) | 8653 (57)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 6250 (5790-6710). | 8999 (49) | 12280 (15) | 13910 (52)

13. Secondary Outcome: Single Dose: Apparent Clearance (CL/F) of PF-06840002 and PF-06840001 [Part 1]
Description: CL/F of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by Dose/Area under the concentration-time profile from time 0 extrapolated to infinite time (AUCinf). The analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: The "Overall Number of Participants Analyzed" represents the total number of participants in the treatment group in the indicated population. The "Number Analyzed" represents the number of participants contributing to the summary statistics, i.e. number of participants where CL/F was determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per minute (mL/min)
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Milliliter per minute (mL/min)
  PF-06840002: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The CL/F of this 1 participant is 527.0 mL/min. | 751.6 (85) |  | 1561 (40)
  PF-06840001: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The CL/F of this 1 participant is 358.0 mL/min. | 454.6 (69) |  | 965.4 (39)

14. Secondary Outcome: Single Dose: Apparent Volume of Distribution (Vz/F) of PF-06840002 and PF-06840001 [Part 1]
Description: Vz/F of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by Dose/(AUC*kel). AUC is the area under concentration curve and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve. The analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: The "Overall Number of Participants Analyzed" represents the total number of participants in the treatment group in the indicated population. The "Number Analyzed" represents the number of participants contributing to the summary statistics, i.e. number of participants where Vz/F was determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Liter
  PF-06840002: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The Vz/F of this 1 participant is 186.0L. | 228.4 (27) |  | 277.2 (20)
  PF-06840001: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The Vz/F of this 1 participant is 97.70L. | 129.3 (12) |  | 159.6 (25)

15. Secondary Outcome: Single Dose: Terminal Half-Life (t1/2) of PF-06840002 and PF-06840001 [Part 1]
Description: t1/2 of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration-time curve. Only those data points judged to describe the terminal log linear decline were used in the regression. The analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: The "Overall Number of Participants Analyzed" represents the total number of participants in the treatment group in the indicated population. The "Number Analyzed" represents the number of participants contributing to the summary statistics, i.e. number of participants where t1/2 was determined.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
hr
  PF-06840002: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840002 | NA (NA) — It is not possible to calculate mean (standard deviation) for insufficient number of participants (n=1), so NA is listed. The t1/2 of this 1 participant is 4.080 hr. | 3.773 (1.5931) |  | 2.090 (0.45033)
  PF-06840001: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840001 | NA (NA) — It is not possible to calculate mean (standard deviation) for insufficient number of participants (n=1), so NA is listed. The t1/2 of this 1 participant is 3.150 hr. | 3.580 (1.5943) |  | 1.943 (0.39273)

16. Secondary Outcome: Single Dose: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06840002 and PF-06840001 [Part 1]
Description: AUCinf of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by AUClast + (Clast/kel), where AUClast is the area under the concentration-time profile from time zero to the time of the last quantifiable concentration, Clast is the predicted serum concentration at the last quantifiable time point estimated from the log linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve. The analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Time Frame: Cycle 1 Day 1 pre-dose, 1, 2, 4, 6, 8, 24 and 72 hours post Cycle 1 Day 1 dose
Population: The "Overall Number of Participants Analyzed" represents the total number of participants in the treatment group in the indicated population. The "Number Analyzed" represents the number of participants contributing to the summary statistics, i.e. number of participants where AUCinf was determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ng*hr/mL
  PF-06840002: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The AUCinf of this 1 participant is 3960 ng*hr/mL. | 5549 (85) |  | 5343 (40)
  PF-06840001: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The AUCinf of this 1 participant is 5820 ng*hr/mL. | 9174 (69) |  | 8645 (39)

17. Secondary Outcome: Multiple Dose: Maximum Observed Plasma Concentration (Cmax) of PF-06840002 and PF-06840001 [Part 1]
Description: Cmax of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) were observed directly from data.
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ng/mL
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 623.0 (463-783). | 779.3 (9) | 1763 (25) | 2474 (66)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 580.5 (468-693). | 1334 (5) | 2810 (24) | 3978 (58)

18. Secondary Outcome: Multiple Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06840002 and PF-06840001 [Part 1]
Description: as for outcome 10
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
hr
  PF-06840002 | 3.00 [2.00 to 4.00] | 3.03 [2.08 to 4.07] | 2.00 [2.00 to 2.10] | 3.02 [1.00 to 4.00]
  PF-06840001 | 3.00 [2.00 to 4.00] | 3.03 [2.08 to 4.07] | 2.00 [2.00 to 2.10] | 3.95 [2.08 to 8.00]

19. Secondary Outcome: Multiple Dose: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06840002 and PF-06840001 [Part 1]
Description: as for outcome 12
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ng*hr/mL
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 6115 (3320-8910). | 6680 (75) | 12730 (50) | 20410 (96)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 10780 (5950-15600). | 10440 (64) | 21020 (50) | 32080 (89)

20. Secondary Outcome: Multiple Dose: Terminal Half-Life (t1/2) of PF-06840002 and PF-06840001 [Part 1]
Description: as for outcome 15
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 15
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
hr
  PF-06840002: number analyzed (Participants) | 2 | 2 | 1 | 2
  PF-06840002 | 5.58 [4.22 to 6.94] | 2.90 [2.16 to 3.64] | 2.68 [2.68 to 2.68] | 2.885 [1.97 to 3.80]
  PF-06840001: number analyzed (Participants) | 2 | 3 | 1 | 2
  PF-06840001 | 5.505 [4.16 to 6.85] | 2.61 [1.92 to 3.63] | 2.50 [2.50 to 2.50] | 2.685 [1.91 to 3.46]

21. Secondary Outcome: Multiple Dose: Lowest Concentration Observed During the Dosing Interval (Cmin) of PF-06840002 and PF-06840001 [Part 1]
Description: Cmin of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was observed directly from data.
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ng/mL
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate mean (standard deviation) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 63.95 (11.9-116). | 15.85 (21.622) | 687.3 (409.76) | 1611 (1749.7)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate mean (standard deviation) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 109.5 (20.9-198). | 21.75 (27.298) | 1079 (587.86) | 2308 (2161.3)

22. Secondary Outcome: Multiple Dose: Average Concentration for the Dosing Interval (Cav) of PF-06840002 and PF-06840001 [Part 1]
Description: Cav of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was observed directly from data.
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ng/mL
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 254.5 (138-371). | 278 (75) | 1060 (50) | 1702 (96)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 449.5 (248-651). | 435.1 (64) | 1755 (49) | 2673 (89)

23. Secondary Outcome: Multiple Dose: Apparent Clearance (CL/F) of PF-06840002 and PF-06840001 [Part 1]
Description: CL/F of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by Dose/Area under the concentration-time profile from time 0 extrapolated to infinite time (AUCinf).
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
mL/min
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 431.0 (234-628). | 624.2 (75) | 327.6 (50) | 408.3 (96)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 241.5 (133-350). | 399.1 (64) | 198.2 (50) | 259.5 (89)

24. Secondary Outcome: Multiple Dose: Apparent Volume of Distribution (Vz/F) of PF-06840002 and PF-06840001 [Part 1]
Description: as for outcome 14
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 14
Measure: Median (Full Range); unit: Liter
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
Liter
  PF-06840002: number analyzed (Participants) | 2 | 2 | 1 | 2
  PF-06840002 | 184.5 [140 to 229] | 216 [202 to 230] | 128 [128 to 128] | 270.5 [269 to 272]
  PF-06840001: number analyzed (Participants) | 2 | 3 | 1 | 2
  PF-06840001 | 102.6 [79.1 to 126] | 117 [114 to 125] | 72.6 [72.6 to 72.6] | 162 [153 to 171]

25. Secondary Outcome: Multiple Dose: Observed Accumulation Ratio (Rac) of PF-06840002 and PF-06840001 [Part 1]
Description: Rac of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by AUCtau (steady state) / AUCtau (single dose).
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ratio
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 1.725 (1.14-2.31). | 1.244 (31) | 1.670 (45) | 2.359 (45)
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=2), so NA is listed. The median (range) was presented for n=2: 1.680 (1.03-2.33). | 1.163 (31) | 1.717 (45) | 2.304 (41)

26. Secondary Outcome: Multiple Dose: Steady State Accumulation Ratio (Rss) of PF-06840002 and PF-06840001 [Part 1]
Description: Rss of PF-06840002 (Active Enantiomer) and PF-06840001 (Inactive Enantiomer) was determined by AUCtau (steady state) / AUCinf (single dose). The analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Time Frame: Cycle 1 Day 15 pre-dose, 1, 2, 4, 6, 8, 24 hrs post
Population: The "Overall Number of Participants Analyzed" represents the total number of participants in the treatment group in the indicated population. The "Number Analyzed" represents the number of participants contributing to the summary statistics, i.e. number of participants where Rss was determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ratio
  PF-06840002: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840002 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The Rss of this 1 participant is 2.250. | 1.289 (37) |  | 1.961 (72)
  PF-06840001: number analyzed (Participants) | 1 | 3 | 0 | 3
  PF-06840001 | NA (NA) — It is not possible and meaningful to calculate geometric mean (geometric CV) for insufficient number of participants (n=1), so NA is listed. The Rss of this 1 participant is 1.020. | 1.266 (31) |  | 1.895 (61)

27. Secondary Outcome: Steady-State Trough Level Ratio [Part 1]
Description: Steady-State trough level ratio was determined by cerebrospinal fluid (CSF)/Plasma. CSF/Plasma ratio was calculated based on the unbound concentration of each analyte. The analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest.
Time Frame: Baseline and Day 15
Population: The "Overall Number of Participants Analyzed" represents the total number of participants in the treatment group in the indicated population. The "Number Analyzed" represents the number of participants contributing to the summary statistics, i.e. number of participants where CSF/Plasma ratio was determined.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ratio
  PF-06840002: number analyzed (Participants) | 0 | 0 | 2 | 4
  PF-06840002 |  |  | 1.00 (0.007) | 1.00 (0.692)
  PF-06840001: number analyzed (Participants) | 0 | 0 | 2 | 4
  PF-06840001 |  |  | 0.89 (0.105) | 0.88 (0.619)

28. Secondary Outcome: Plasma Kynurenine and Tryptophan [Part 1]
Description: The levels of Kynurenine and Tryptophan in blood samples were determined using the qualified analytical method.
Time Frame: Cycle 1 Day 1 pre-dose, and 1, 2, 4, 6, 8, 24 hours post-dose; Cycle 1 Day 4 and Day 8 pre-dose; Cycle 1 Day 15 pre-dose, and 1, 2, 4, 6, 8, 24 hours post-dose
Population: The analysis population was the total number of participants in the treatment group in the indicated population.
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
micromolar
  Kynurenine | 1.545 (0.2051) | 2.185 (1.7443) | 1.144 (0.1479) | 1.523 (0.4321)
  Tryptophan | 48.15 (4.596) | 29.55 (4.611) | 36.77 (7.681) | 33.10 (4.590)

29. Secondary Outcome: Plasma Endogenous Kynurenine/Tryptophan Ratio [Part 1]
Description: The Kynurenine/Tryptophan ratio was determined by 1000*Kynurenine/Tryptophan.
Time Frame: as for outcome 28
Population: The "Number of Participants Analyzed" represents the total number of participants in the treatment group in the indicated population on Cycle 1 Day. The "Number Analyzed" represents the number of participants contributing to the summary statistics at the end of treatment.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
Number analyzed (Participants) | 2 | 4 | 3 | 8
ratio | 38.467 (0.6791) | 53.066 (24.9722) | 25.854 (7.6209) | 42.463 (NA) — The number of participants in the group "PF-06840003 500 MG BID" on Cycle 1 Day 1 was 8 but the number of participants analyzed at the end of treatment was n=1. It is not possible to calculate standard deviation for n=1, therefore NA was listed.

ADVERSE EVENTS:
Time Frame: Baseline up to 1 year
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | PF-06840003 125 MG QD | PF-06840003 250 MG QD | PF-06840003 250 MG BID | PF-06840003 500 MG BID
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 0/3 | 3/8
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06840003 125 MG QD (N=2) | PF-06840003 250 MG QD (N=4) | PF-06840003 250 MG BID (N=3) | PF-06840003 500 MG BID (N=8)
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06840003 125 MG QD (N=2) | PF-06840003 250 MG QD (N=4) | PF-06840003 250 MG BID (N=3) | PF-06840003 500 MG BID (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 3
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 3 | 1 | 4
Influenza like illness (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Protein total increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 4
Apraxia (Nervous system disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 2
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 2
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 2 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Visual field defect (Nervous system disorders) | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Part 2 of the study was not initiated. Because after reviewing efficacy, safety, PK and PD of all available data from enrolled patients, the Sponsor decided to prematurely terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02764151/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT02764151/SAP_001.pdf